CLINICAL TRIAL: NCT05071365
Title: Early Access to Virtual Resources for the Self-management of Plantar Fasciitis: A Proof of Concept and Feasibility Study
Brief Title: Early Access to Virtual Resources for the Self-management of Plantar Fasciitis
Acronym: EASE-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8125
Record Dates: First submitted 2021-08-03; First posted 2021-10-08 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-03

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Videos (Experimental): Single Arm study: All participants recruited to the study will be allocated to a single arm- "videos" in which participants will be able to access self help videos for plantar fasciitis
  Interventions: Other: Early access to virtual resources

INTERVENTIONS:
Other: Early access to virtual resources — Single arm study. Participants are given access to self help videos for the management of plantar fasciitis while they are on the waiting list

SUMMARY:
This proof of concept and feasibility study will adopt a mixed methods approach. The primary objectives will be to assess participants' acceptance and usability of a package of self-help videos for Plantar Fasciitis designed to be accessed shortly after suitable participants are referred to the podiatry service, and also the feasibility of conducting a future randomised controlled trial. The secondary objectives will be to assess the effects of the intervention on pain and quality of life.

DETAILED DESCRIPTION:
This proof of concept and feasibility project will investigate the use of a self-help package of virtual resources for the treatment of plantar fasciitis. The research will involve a small group of ten, shortly after participants are referred to Cardiff & Vale UHB podiatry service and join the waiting list.

The virtual resources will include short videos demonstrating ways of managing symptoms, such as gentle stretching exercises, and footwear recommendations. Participants will be given access to these resources to watch at their convenience. Patient reported outcome measures (foot pain, and quality of life) will be collated at baseline and periodically up to 6 weeks. Participants' acceptability of these resources will be assessed through interviews at the end of the six weeks.

The feasibility of conducting a future randomised controlled trial will be assessed by looking at recruitment rates, retention and any patient safety issues. It is hoped the long term benefit will be that participants joining the waiting list can engage with these resources at the earliest opportunity to help manage their symptoms.

This research is important because it presents an opportunity to work with participants at the start of joining a waiting list, and the benefits of early access to virtual resources could be applicable to a number of different health problems.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

* Diagnosis of Plantar Fasciitis by assessing podiatrist:
* Plantar medial heel pain: most noticeable with initial steps after a period of inactivity (post static dyskinesia) but also worse following prolonged weight bearing
* Pain with palpation of the proximal insertion of the plantar fascia, most commonly the medial calcaneal tubercle, the site of the plantar aponeurosis (Clinical pressure application to locate the most tender spot in order to anatomically describe the site).
* Symptomatic for PF for any time period
* ≥18 years of age
* Able to provide informed consent
* Access to internet

Exclusion Criteria:

* Diabetes or neuropathy
* History of systemic diseases such as inflammatory joint disease, rheumatic, autoimmune or neurological conditions.
* Chronic pain syndrome or lumbosacral radiculitis
* Pregnancy
* Orthopaedic surgery (spinal/ lower limb within the last year)
* Corticosteroid injection for plantar fasciitis in the last 6 months (prior to onset)
* Plantar heel pain related to fractures, tumours, infection, nerve entrapment or in the opinion of the assessing podiatrist confounded by any other medical condition
* Patient unable to complete exercises in self-help resources
* Unable to access internet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Acceptability of resources as assessed through semi structured interviews | 6 weeks
  End of study semi-structured interviews, analysed using a thematic approach.
Usability of resources as assessed through semi structured interviews | 6 weeks
  End of study semi-structured interviews, analysed using a thematic approach
Feasibility as assessed through recruitment and retention rates | 6 weeks
  End of study assessment of feasibility through recruitment and retention rates.
Feasibility as assessed through adverse events. | 6 weeks
  End of study assessment of feasibility through adverse events

SECONDARY OUTCOMES:
Assess effects of intervention on pain using Visual Analogue Scale with higher scores indicating a worse outcome | 6 weeks
  Patient reported outcome measures recorded at baseline, 2 4 and 6 weeks
Assess effects of intervention on quality of life using EQ5D (EuroQol) with higher scores indicating a worse outcome | 6 weeks
  Patient reported outcome measures at baseline, 2 4 and 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical research facility, Cardiff, United Kingdom